CLINICAL TRIAL: NCT00309686
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Flexibly-Dosed Extended-Release Paliperidone as Adjunctive Therapy to Mood Stabilizers in the Treatment of Acute Manic and Mixed Episodes Associated With Bipolar I Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Adjustable Doses of Extended-release (ER) Paliperidone Compared With Placebo, in Combination With Lithium or Valproate, to Treat Manic and Mixed Episodes in Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR010855
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-03

CONDITIONS: Affective Psychosis, Bipolar; Bipolar Disorder; Mania
Keywords: Affective psychosis; bipolar disorder; manic disorder; manic-depressive psychosis; mania; manic state; paliperidone; paliperidone ER; adjunctive therapy
MeSH Terms: conditions — Bipolar Disorder; Mania; Affective Disorders, Psychotic | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety over a 6-week period of paliperidone ER compared with placebo in treating subjects with Bipolar I Disorder who are experiencing a manic or mixed episode while they are taking lithium or valproate. This study will also evaluate the effect of paliperidone ER compared with placebo on overall functioning, on how quickly a response is seen, on improvement in severity of illness, on health-related functional status, on depressive symptoms, and on psychotic symptoms. The relationship between blood levels and the effectiveness and safety of paliperidone ER will be evaluated, including the effect of food relative to time of taking the drug.

DETAILED DESCRIPTION:
Several treatments are available for the treatment of acute manic and mixed episodes associated with bipolar disorder. Some of these treatments, including lithium, divalproex sodium, and carbamazepine, have been used for many years. More recently, risperidone and a number of atypical antipsychotics (olanzapine, quetiapine, ziprasidone, aripiprazole) have been approved for use in the treatment of acute mania. Paliperidone has similar properties to risperidone and is thus expected to have at least similar efficacy to risperidone in the treatment of acute manic and mixed episodes associated with bipolar disorder. Paliperidone ER has been shown to be effective in treating schizophrenia, and has an improved delivery system (with delivery at a relatively controlled rate over 24 hours) and a reduced potential for drug-drug interactions. Treatment of bipolar mania often involves more than a single medication. Studies of mood stabilizers in combination with antipsychotic agents have suggested greater efficacy or more rapid onset of action with these combinations than with any of these agents alone. It is therefore of interest to evaluate the effectiveness of paliperidone ER in combination with mood stabilizers for the treatment of acute manic and mixed episodes associated with bipolar disorder.

This randomized (patients are randomly assigned to receive paliperidone ER or placebo), double-blind (neither the patient nor the physician knows whether drug or placebo and what dosage is being taken), placebo-controlled, parallel-group, multicenter study will evaluate paliperidone ER compared with placebo over a 6-week period in patients with Bipolar I Disorder who are experiencing an acute manic or mixed episode and are taking lithium or valproate. A flexible dosing regimen will be used in this study to afford investigators the ability to adjust the dosage of each subject to achieve rapid control of acute manic symptoms. After a screening/washout phase of no more than 7 days to determine if patients are eligible and to discontinue all medications excluded per protocol criteria(including any mood-stabilizing medications other than lithium or valproate), patients will be randomly assigned to either paliperidone ER or placebo for a 6-week, double-blind treatment phase. Patients will be hospitalized for at least the first 7 days, and will be discharged and followed as outpatients only if they are considered to be at no significant risk of violent or suicidal behavior. An end-of-study visit will be conducted at the end of the double-blind treatment phase or at early withdrawal, whichever comes first. A follow-up (post-treatment) visit for safety evaluations will be scheduled approximately 1 week after the end-of-study/early withdrawal visit. The study, including the screening/washout phase, will last up to 56 days (8 weeks).

Effectiveness will primarily be determined by the change from baseline in the Young Mania Rating Scale (YMRS) score to the end of the 6-week double-blind treatment phase or early withdrawal. The YMRS is an established 11-item scale used to evaluate manic symptoms. A secondary measure of effectiveness will be the change from baseline in the Global Assessment of Functioning (GAF) score to the end of the 6 weeks of treatment. Additional measures of effectiveness will measure severity of bipolar illness, psychotic symptoms, quality of sleep, and health-related functional status. Safety will be measured by monitoring the frequency, severity, and timing of side effects; monitoring the need for additional medications; clinical laboratory tests (including pregnancy tests), 12-lead electrocardiograms; measurement of vital signs (blood pressure, pulse, and temperature); and physical examination (including height, weight, and waist circumference). Three scales will be used to assess specific neurologic side effects; the Scale for Suicidal Ideation will be used to evaluate any suicidal tendencies. The primary study hypothesis is that, in the treatment of patients who experience an acute manic or mixed episode while they are taking lithium or valproate for the treatment of Bipolar I Disorder, paliperidone ER is superior to placebo on the change from baseline in the YMRS total score at the end of 6 weeks of double-blind treatment. The secondary hypothesis is that, in these same patients, paliperidone ER is superior to placebo on the change from baseline in GAF score at the end of 6 weeks of double-blind treatment. Flexibly dosed oral paliperidone ER (3 to 12 mg/day) or matching placebo once daily. All study drug will be administered before 10:00 a.m. Initial dosage will be 6 mg/day; adjustment of the dosage will be based on assessment of the patient's response to and tolerance of the study drug. Dosage may be increased in 3-mg/day increments or decreased as deemed necessary; dosage should only be increased every 2 days unless a patient requires a higher dosage to control manic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV) criteria for Bipolar I Disorder, Most Recent Episode Manic or Mixed (with or without psychotic features)
* History of at least 1 previously documented manic or mixed episode requiring medical treatment within the past 3 years
* Must have been taking lithium or valproate as part of treatment for Bipolar I Disorder for at least 2 weeks before screening, with drug levels at screening within therapeutic range
* Total YMRS score of at least 20 at screening and at baseline (Day 1)
* Women must be postmenopausal for at least 2 years or agree to practice an effective method of birth control throughout the study.

Exclusion Criteria:

* Meets DSM-IV criteria for rapid cycling and schizoaffective disorder
* In the opinion of the study doctor, is at significant risk for suicidal or violent behavior during the course of the study
* Has used cocaine, phencyclidine, amphetamine, methylphenidate, pemoline, an opioid (excluding codeine), hallucinogen, or any other drug that may be associated with manic symptoms as evidenced by a positive urine drug screen
* Has received benzodiazepines at doses equal to 4 mg/day of lorazepam or higher for a period of 3 months or longer immediately before the screening phase.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness outcome is the change in total YMRS score from baseline (first dose) to the last assessment in the 6-week double-blind treatment phase.

SECONDARY OUTCOMES:
The secondary effectiveness outcome is the change in GAF score from baseline (first dose) to the last assessment in the 6-week double-blind treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Berwaerts J, Lane R, Nuamah IF, Lim P, Remmerie B, Hough DW. Paliperidone extended-release as adjunctive therapy to lithium or valproate in the treatment of acute mania: a randomized, placebo-controlled study. J Affect Disord. 2011 Mar;129(1-3):252-60. doi: 10.1016/j.jad.2010.09.011. Epub 2010 Oct 13. PMID 20947174
- See also: A Study to Evaluate the Efficacy and Safety of Adjustable Doses of Extended-Release (ER) Paliperidone Compared With Placebo, in Combination With Lithium or Valproate, to Treat Manic and Mixed Episodes in Patients With Bipolar I Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=721&filename=CR010855_CSR.pdf